CLINICAL TRIAL: NCT01094639
Title: Periodontal Infection and Systemic Inflammation in Renal Patients
Acronym: PeriRen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Efthimia Ioannidou, Associate Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-092-2; K23DE018689 (NIH)
Record Dates: First submitted 2010-03-23; First posted 2010-03-29 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Periodontitis; Chronic Kidney Disease
MeSH Terms: conditions — Periodontitis; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supragingival prophylaxis (Placebo Comparator): Plaque removal
  Interventions: Procedure: Supragingival Prophylaxis
- Scaling root planing (Active Comparator): SRP+oral hygiene
  Interventions: Procedure: Scaling root planing

INTERVENTIONS:
Procedure: Scaling root planing — Deep gum cleaning with local anesthesia
  Arms: Scaling root planing
Procedure: Supragingival Prophylaxis — Plaque removal
  Arms: Supragingival prophylaxis

SUMMARY:
The purpose of this study is to examine the role of gum disease in affecting the long term prognosis of renal patients. This disease if untreated causes inflammatory response throughout the body. If the subject has gum disease, he/she will be randomly assigned to one of the two treatment groups. The study investigates what happens to inflammatory markers in blood and saliva after you are treated for gum disease.

DETAILED DESCRIPTION:
The main goal of this project was to explore the contribution of chronic periodontitis to systemic inflammation in Chronic Kidney Disease (CKD). To achieve this goal, the project had two specific objectives:

1. a) To compare the prevalence of periodontal infection between CKD and non-CKD populations and b) to explore the association between the presence of periodontal infection and the uremic status of CKD patients.
2. a) To assess the levels of systemic inflammatory markers, IL-6 and CRP in the presence or absence of periodontal infection in CKD and b) to compare the serum IL-6 and CRP levels in response to periodontal intervention.

ELIGIBILITY:
Inclusion Criteria:

* dental subjects with periodontitis,
* at least 10 teeth
* no periodontal (gum) treatment for the last year,
* no antibiotic for the last 4 months,
* no vascular access infection.

Exclusion Criteria:

* smokers

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-08; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Serum Interleukin-6 (IL-6) and C-reactive protein (CRP) levels | 2 months
  IL-6 and CRP are markers of systemic inflammation and may improve at the end of gum treatment.

SECONDARY OUTCOMES:
Changes in periodontal (gum) clinical presentation and status | 2 months
  For the secondary outcome, periodontal variables such as bleeding on probing, probing depth (the depth of the gum sulcus around the tooth), and bacterial plaque score will be evaluated to assess the effectiveness of the intervention and the compliance of the patients

CONTACTS AND LOCATIONS:
Overall Officials: Efthimia Ioannidou, DDS, MDS, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ioannidou E, Malekzadeh T, Dongari-Bagtzoglou A. Effect of periodontal treatment on serum C-reactive protein levels: a systematic review and meta-analysis. J Periodontol. 2006 Oct;77(10):1635-42. doi: 10.1902/jop.2006.050443. PMID 17032104
- [Background] Ioannidou E, Shaqman M, Burleson J, Dongari-Bagtzoglou A. Periodontitis case definition affects the association with renal function in kidney transplant recipients. Oral Dis. 2010 Oct;16(7):636-42. doi: 10.1111/j.1601-0825.2010.01665.x. PMID 20412451
- [Background] Ioannidou E, Swede H, Dongari-Bagtzoglou A. Periodontitis predicts elevated C-reactive protein levels in chronic kidney disease. J Dent Res. 2011 Dec;90(12):1411-5. doi: 10.1177/0022034511423394. Epub 2011 Sep 22. PMID 21940520
- [Background] Hong BY, Furtado Araujo MV, Strausbaugh LD, Terzi E, Ioannidou E, Diaz PI. Microbiome profiles in periodontitis in relation to host and disease characteristics. PLoS One. 2015 May 18;10(5):e0127077. doi: 10.1371/journal.pone.0127077. eCollection 2015. PMID 25984952
- [Result] Ioannidou E, Swede H. Disparities in periodontitis prevalence among chronic kidney disease patients. J Dent Res. 2011 Jun;90(6):730-4. doi: 10.1177/0022034511402209. Epub 2011 Mar 21. PMID 21422478
- [Result] Ioannidou E, Hall Y, Swede H, Himmelfarb J. Periodontitis associated with chronic kidney disease among Mexican Americans. J Public Health Dent. 2013 Spring;73(2):112-9. doi: 10.1111/j.1752-7325.2012.00350.x. Epub 2012 Jul 6. PMID 22775287
- [Result] Araujo MV, Hong BY, Fava PL, Khan S, Burleson JA, Fares G, Samson W, Strausbaugh LD, Diaz PI, Ioannidou E. End stage renal disease as a modifier of the periodontal microbiome. BMC Nephrol. 2015 Jun 9;16:80. doi: 10.1186/s12882-015-0081-x. PMID 26055269
- [Result] Ioannidou E, Swede H, Fares G, Himmelfarb J. Tooth loss strongly associates with malnutrition in chronic kidney disease. J Periodontol. 2014 Jul;85(7):899-907. doi: 10.1902/jop.2013.130347. Epub 2013 Nov 11. PMID 24215204